CLINICAL TRIAL: NCT00137462
Title: A Phase 3, Double-Blind, Randomized, Multisite Trial Of The Efficacy, Safety, And Tolerability Of The Fixed Combination Torcetrapib/Atorvastatin Administered Orally, Once Daily For 12 Months, Compared To Atorvastatin Alone, Titrated Based On NCEP ATP-III LDL-C Goals In Subjects With Fredrickson Types IIa And IIb Dyslipidemias
Brief Title: Lipitor Trial To Study The Effect Of Torcetrpib/Atorvastatin To Atorvastatin Alone.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5091019
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2006-12

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — torcetrapib; Atorvastatin

INTERVENTIONS:
Drug: torcetrapib/atorvastatin
Drug: atorvastatin

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

To look at various lipids in the blood of people with Fredrickson Type IIa and Type IIb mixed dyslipidemias

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* Statin eligible per NCEP ATP-III guidelines
* At least 18 years of age

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant
* Intolerance to statin therapy
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluation of response, or render unlikely that the subject would complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2004-11; Study Completion 2006-09

PRIMARY OUTCOMES:
Change in lipid parameters (HDL, LDL) at various timepoints over 12 months.

SECONDARY OUTCOMES:
Changes in levels of lipids and other biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (43):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Union Grove, Alabama
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Golden, Colorado
  - Pfizer Investigational Site, Bridgeport, Connecticut
  - Pfizer Investigational Site, Fairfield, Connecticut
  - Pfizer Investigational Site, Trumbull, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Boynton Beach, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Gainsville, Florida
  - Pfizer Investigational Site, Sebastian, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Olathe, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Burlington, Massachusetts
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Orchard Park, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Keizer, Oregon
  - Pfizer Investigational Site, Salem, Oregon
  - Pfizer Investigational Site, Doylestown, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Morristown, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, McKinney, Texas
- Canada (10):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Charlottetown, Prince Edward Island
  - Pfizer Investigational Site, Mirabel, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Saint Georges de Beauce, Quebec